CLINICAL TRIAL: NCT00340977
Title: Svangerskap, Arv, Og Miljo (Pregnancy, Heredity and Environment)
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996006; OH96-E-N006
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11-18

CONDITIONS: Birth Defects; Cleft Palate; Cleft Lip
Keywords: Birth Defects; Cleft Lip and Palate; Genetic Susceptibility
MeSH Terms: conditions — Congenital Abnormalities; Cleft Palate; Cleft Lip; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Case-Control Parent-Triad: Norwegian infants born with cleft lip or palate over a 5 year period

SUMMARY:
This proposal describes a population-based case-control study of all Norwegian infants born with cleft lip or palate over a five-year period. The study will be jointly supported by the U.S. National Institute of Environmental Health Sciences (NIEHS), and the Norwegian National Institute of Public Health (SIFF) and Medical Birth Registry of Norway (MBR). Cases will be identified through the two surgery clinics that treat all clefts in Norway. Controls will be randomly selected from all live births through the MBR. Mothers will complete two selfadministered questionnaires; one regarding exposures before and during pregnancy, the other their diet during their early months of pregnancy. Biological specimens for DNA testing (blood samples, buccal swabs) will be collected from cases, controls and mothers in order to describe possible gene-environment interactions. With 750 cases and 1100 controls, this will be one of the largest and most complete field studies of facial clefting yet conducted.

DETAILED DESCRIPTION:
This proposal describes a population-based case-control study of all Norwegian infants born with cleft lip or palate over a five-year period. The study will be jointly supported by the U.S. National Institute of Environmental Health Sciences (NIEHS), and the Norwegian National Institute of Public Health (SIFF) and Medical Birth Registry of Norway (MBR). Cases will be identified through the two surgery clinics that treat all clefts in Norway. Controls will be randomly selected from all live births through the MBR. Mothers will complete two selfadministered questionnaires; one regarding exposures before and during pregnancy, the other their diet during their early months of pregnancy. Biological specimens for DNA testing (blood samples, buccal swabs) will be collected from cases, controls and mothers in order to describe possible gene-environment interactions. With 750 cases and 1100 controls, this will be one of the largest and most complete field studies of facial clefting yet conducted.

ELIGIBILITY:
* INCLUSION CRITERIA:

We expect to enroll about 150 infants with cleft lip or palate annually for five years (550 with cleft lip with or without cleft palate, and 200 with cleft palate alone)

Controls will be chosen randomly from all Norwegian live-births through the Medical Birth Registry.

EXCLUSION CRITERIA:

There will be no exclusion by race, sex or ethnic group.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4091 (Actual)
Dates: Start 1995-09-06; Study Completion 2019-11-18

PRIMARY OUTCOMES:
Identification of genetic alleles | Ascertained within first year after birth
  Facial Clefts

CONTACTS AND LOCATIONS:
Overall Officials: Allen Wilcox, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- Norway (2):
  - Norwegian Institute of Public Health, Bergen
  - University of Bergen, Bergen

REFERENCES:
- [Background] Abyholm FE, Borchgrevink HC, Eskeland G. Cleft lip and palate in Norway. III. Surgical treatment of CLP patients in Oslo 1954-75. Scand J Plast Reconstr Surg. 1981;15(1):15-28. doi: 10.3109/02844318109103407. No abstract available. PMID 7268309
- [Background] Abyholm FE. Cleft lip and palate in a Norwegian population. II. A numerical study of 1555 CLP-patients admitted for surgical treatment 1954-75. Scand J Plast Reconstr Surg. 1978;12(1):35-43. doi: 10.3109/02844317809010478. No abstract available. PMID 663563
- [Background] Abyholm FE. Cleft lip and palate in Norway. I. Registration, incidence and early mortality of infants with CLP. Scand J Plast Reconstr Surg. 1978;12(1):29-34. doi: 10.3109/02844317809010477. No abstract available. PMID 566463